CLINICAL TRIAL: NCT04597203
Title: Efficacy and Safety of Using Combination of 755-nm Picosecond Alexandrite Laser and 2% Hydroquinone Compared With 2% Hydroquinone Alone for the Treatment of Melasma: a Randomized Split-face Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: si 082/2019
Record Dates: First submitted 2020-09-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — hydroquinone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- split face - left side (Experimental)
  Interventions: Device: 755-nm picosecond alexandrite laser with topical 2% hydroquinone
- split face - right side (Active Comparator)
  Interventions: Drug: topical 2% hydroquinone

INTERVENTIONS:
Device: 755-nm picosecond alexandrite laser with topical 2% hydroquinone — treatment one side of the face with 755-nm picosecond alexandrite laser with topical 2% hydroquinone
  Arms: split face - left side
Drug: topical 2% hydroquinone — treatment one side of the face with topical 2% hydroquinone
  Arms: split face - right side

SUMMARY:
This study aims to assess the efficacy and safety of using combination of 755-nm picosecond alexandrite laser and 2% hydroquinone compared with 2% hydroquinone alone for the treatment of melasma: A randomized split-face controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Both male and female age 18-60 years
* Melasma on both cheeks - epidermal or mixed type
* Fitzpatrick Skin type III-V

Exclusion Criteria:

* History of retinoid or other keratolytic drugs used within 6 months before enrolled
* History of keloid
* photosensitivity
* Immunocompromised host

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Modified melasma area and severity index score(mMASI) - comparing between Picosecond laser 755 nm with 2%HQ and 2%HQ alone for treatment of melasma of using combination of 755-nm picosecond alexandrite laser and 2% hydroquinone | 6 months
  score range 0-24
Melanin index measured by Mexameter® - comparing between Picosecond laser 755 nm with 2%HQ and 2%HQ alone for treatment of melasma | 6 months
  measuring in au
Average melanin measured by Antera3D® - comparing between Picosecond laser 755 nm with 2%HQ and 2%HQ alone for treatment of melasma | 6 months
  measuring in au
Patient satisfaction quartile score - comparing between Picosecond laser 755 nm with 2%HQ and 2%HQ alone for treatment of melasma | 6 months
  score 0 -100%
Physician evaluation quartile score - comparing between Picosecond laser 755 nm with 2%HQ and 2%HQ alone for treatment of melasma | 6 months
  score 0 -100%

SECONDARY OUTCOMES:
Safety of using combination of 755-nm picosecond alexandrite laser | 6 months
  Monitor side effect from picesecond alexandrite laser
Safety of using 2% hydroquinone | 6 months
  side effect of topical 2%Hydroquinone use

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manuskiatti W, Yan C, Gulfan MCB, Techapichetvanich T, Wanitphakdeedecha R. Combination of a 755-nm picosecond laser and hydroquinone 2% cream versus hydroquinone 2% cream alone for the treatment of melasma: A randomized, split-face, and controlled trial. Lasers Surg Med. 2022 Dec;54(10):1245-1250. doi: 10.1002/lsm.23615. Epub 2022 Nov 8. PMID 36345697